CLINICAL TRIAL: NCT00029861
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dose, Multicenter Study of Weight-Reducing and Prevention of Weight Regain Effects and Safety in Obese Patients With or Without Comorbidities
Brief Title: Obese Patients With or Without Comorbidities (RIO-North America)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFC4743
Record Dates: First submitted 2002-01-23; First posted 2002-01-24 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Obesity; Weight Loss
Keywords: Weight Loss; Obesity; Weight Reduction; Overweight
MeSH Terms: conditions — Obesity; Weight Loss; Overweight | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Rimonabant (SR141716)

SUMMARY:
To assess the effects of weight loss and weight maintenance over a period of two years when prescribed with a hypocaloric diet in obese patients with or without comorbidities

ELIGIBILITY:
* Stable weight (variation of less than 5 kg within 3 months prior to screening visit)
* BMI (Body Mass Index) of 30 or greater in patients with or without comorbidities, or BMI greater than 27 in patients with treated or untreated hypertension and/or treated or untreated dyslipidemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3045 (Actual)
Dates: Start 2001-08; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Change in body weight

SECONDARY OUTCOMES:
Metabolic parameters

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (51):
- United States (47):
  - Radiant Research, Birmingham, Alabama
  - Radiant Research, Phoenix, Arizona
  - East Bay Clinical Trial Center, Concord, California
  - Feighner Research Institute, San Diego, California
  - Scripps Clinic, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Ranch View Family Medicine, Highlands Ranch, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - Health Core, Inc., Newark, Delaware
  - George Washington Univ. Wieght Mmgt Program, Washington D.C., District of Columbia
  - Miami Research Associates, Miami, Florida
  - Anchor Research Center, Naples, Florida
  - Central Florida Clinical Solutions, Ocoee, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Medical Dietetics, Inc., Atlanta, Georgia
  - Springfield Diabetes and Endocrine Center, Springfield, Illinois
  - Medical Research Consortium, Indianapolis, Indiana
  - Wichita Clinic, PA, Wichita, Kansas
  - University of KY Internal Medicine, Lexington, Kentucky
  - Pennington Center, Baton Rouge, Louisiana
  - JM Clinical Trials, Inc., Swansea, Massachusetts
  - Montana Medical Research, LLC, Missoula, Montana
  - Endocrinology and Diabetes Consultants, PC, Dover, New Hampshire
  - Radiant Research, Lawrenceville, New Jersey
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Central New York Clinical Research, Manlius, New York
  - Comprehensive Weight Control Program, New York, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - Center for Nutrition and Preventive Medicine, Charlotte, North Carolina
  - Multi-Specialty Research Associates of North Carolina, Raleigh, North Carolina
  - South Dayton Research Associates, Beavercreek, Ohio
  - Lindner Clinical Trials Center, Cincinnati, Ohio
  - Radiant Research, Columbus, Ohio
  - Radiant Research, Portland, Oregon
  - SFM Clinical Trials, Scotland, Pennsylvania
  - Radiant Research, Wyomissing, Pennsylvania
  - ClinSearch, Chattanooga, Tennessee
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - Radiant Research, Austin, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - nTouch Research, Houston, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Advanced Clinical Research, Salt Lake City, Utah
  - Commonwealth Clinical Research Specialists (CCRS), Richmond, Virginia
  - Rainer Clinical Research Center, Inc., Renton, Washington
  - Clinical Nutrition Clinic, University of Wisconsin, Madison, Wisconsin
- Canada (4):
  - Corunna Medical Clinic, Corunna, Ontario
  - Quarry Family Medicine Clinic, Kingston, Ontario
  - Trial Management Group, Richmond Hill, Ontario
  - Group North, Windsor, Ontario

REFERENCES:
- [Result] Pi-Sunyer FX, Aronne LJ, Heshmati HM, Devin J, Rosenstock J; RIO-North America Study Group. Effect of rimonabant, a cannabinoid-1 receptor blocker, on weight and cardiometabolic risk factors in overweight or obese patients: RIO-North America: a randomized controlled trial. JAMA. 2006 Feb 15;295(7):761-75. doi: 10.1001/jama.295.7.761. PMID 16478899